CLINICAL TRIAL: NCT01855100
Title: Belgian Real Life Non-interventional Study (NIS) in Patients Treated With Xarelto® Following an Acute Deep Vein Thrombosis (DVT)
Brief Title: Belgian Real Life Non-interventional Study (NIS) in Patients Treated With Xarelto Following an Acute Deep Vein Thrombosis (DVT)
Acronym: BOX-DVT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16852; XA1314BE (Other: Company internal)
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thrombosis
Keywords: Treatment of acute deep vein thrombosis; Prevention of recurrence; Oral anticoagulation; Real-life setting
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Starting dose (3 weeks): 15 mg BID, then 15 mg OD or 20 mg OD.

SUMMARY:
The objective of this NIS is to assess in a real-life setting, usage patterns and associated outcomes in the management (healthcare resource utilisation and associated costs) of patients with acute deep vein thrombosis treated with Xarelto, in accordance with the terms of the European marketing authorization and the Belgian reimbursement criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of deep vein thrombosis (DVT) within the past 9 months, enabling at least 3 months of therapy

Exclusion Criteria:

* Patients who do not fulfil the Belgian reimbursement criteria of deep vein thrombosis (DVT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory or hospitalized patients coming from the vascular diseases clinic of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with major bleedings | up to 1 year or 30 days after end of rivaroxaban
Number of patients with symptomatic recurrent Venous Thrombus Embolism (VTE) | up to 1 year or 30 days after end of rivaroxaban
All-cause mortality | up to 1 year or 30 days after end of rivaroxaban
Adverse events | up to 1 year or 30 days after end of rivaroxaban
Treatment satisfaction measured by means of Anti-clot treatment scale (ACTS) | up to 1 year or 30 days after end of rivaroxaban
Quantities of resource use consumption | up to 1 year or 30 days after end of rivaroxaban

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Belgium